CLINICAL TRIAL: NCT03778424
Title: An Extended Access Program (EAP) for Rufinamide in Pediatric Participants With Inadequately Controlled Lennox-Gastaut Syndrome
Brief Title: An Extended Access Program (EAP) for Participants Who Have Completed Rufinamide Study E2080-G000-303
Status: Available | Type: Expanded Access
Sponsor: Eisai Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: E2080-E044-501
Record Dates: First submitted 2018-11-27; First posted 2018-12-19 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Lennox Gastaut Syndrome
Keywords: Central Nervous System; E2080; Rufinamide; Epilepsy; Seizures; Brain Diseases
MeSH Terms: conditions — Lennox Gastaut Syndrome; Epilepsy; Seizures; Brain Diseases | interventions — rufinamide

STUDY DESIGN:
Expanded Access Types: Individual, Treatment

INTERVENTIONS:
Drug: Rufinamide — Rufinamide up to 45 milligram per kilogram per day (mg/kg/day).

SUMMARY:
This is an extended access study for participants who have completed Rufinamide Study E2080-G000-303 to continue to have access to rufinamide until it becomes commercially available in Poland or until no participants remain in the EAP.

ELIGIBILITY:
Inclusion Criteria:

* Participants who were on rufinamide treatment and have completed Study E2080-G000-303 in Poland.

Exclusion Criteria:

* Participants were randomized to the other antiepileptic drug (AED) treatment group in study E2080-G000-303.

Min Age: 4 Years | Sex: All
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (2):
- Poland (2):
  - Generała Tadeusza Kościuszki 52, Kielce
  - Szpital Kliniczny im. Heliodora Święcickiego Uniwersytetu Medycznego im. Karola Marcinkowskiego w Poznaniu, Poznan